CLINICAL TRIAL: NCT01253642
Title: A Phase II Study of MAOA Inhibitor Plus Docetaxel in Patients Receiving and Progressing on Docetaxel Therapy
Brief Title: Phenelzine Sulfate and Docetaxel in Treating Patients With Prostate Cancer With Progressive Disease After First-Line Therapy With Docetaxel
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); The Wayne D. Kuni and Joan E. Kuni Foundation (Other)
Responsible Party: Principal Investigator, Tom Beer, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00005688; NCI-2010-02037 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SOL-09105-LM; 5688; OHSU-5688; e5688; MR00045508; MR46390; IRB00005688 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2010-11-15; First posted 2010-12-03 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Prostatic Adenocarcinoma; Prostate Adenocarcinoma; Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Phenelzine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (antiangiogenesis, chemosensitizer, chemotherapy) (Experimental): Patients receive phenelzine sulfate PO QD on days -7 to -4, and then BID on days -3 to 21. Patients receive docetaxel IV over 60 minutes on day 1. Treatment repeats every 21 days for at least 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy of Prostate; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Drug: Phenelzine Sulfate

INTERVENTIONS:
Procedure: Biopsy of Prostate — Undergo transrectal ultrasound (TRUS) guided prostate biopsy OR image-guided (CT or ultrasound) core bone or soft tissue biopsy
  Other Names: Prostate Biopsy; Prostatic Biopsy
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Phenelzine Sulfate — Given PO
  Other Names: Nardil

SUMMARY:
This phase II trial studies how well giving phenelzine sulfate together with docetaxel works in treating patients with prostate cancer that is growing, spreading, or getting worse after first-line therapy with docetaxel. Phenelzine sulfate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Phenelzine sulfate may also help docetaxel work better by making tumor cells more sensitive to the drug. Giving phenelzine sulfate together with docetaxel may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the proportion of patients who experience a prostate specific antigen (PSA) decline of at least 30% within 12 weeks of initiation of combination therapy when phenelzine (phenelzine sulfate) is added to docetaxel in patients who have evidence of progression on standard docetaxel.

SECONDARY OBJECTIVES:

I. To determine duration of progression free survival after initiation of combination phenelzine and docetaxel therapy.

II. To determine the response rate in measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria after initiation of combination phenelzine and docetaxel therapy.

III. To report the maximum change in PSA from baseline to 12 weeks (or earlier in patients who discontinue early) by waterfall plot after initiation of combination phenelzine and docetaxel therapy.

IV. To determine the toxicity of the combination regimen in castration-resistant prostate cancer (CRPC) previously treated with docetaxel.

V. To determine time to death from all causes. VI. To determine the frequency of monoamine oxidase A (MAOA) overexpression in CRPC tumors that are progressing on docetaxel.

VII. To compare the level of MAOA expression in primary diagnostic tissue (e.g. biopsy or radical prostatectomy) with CRPC tumors that are progressing on docetaxel.

VIII. To correlate MAOA overexpression in CRPC tumors with response to combination study treatment.

IX. To collect blood and tissue specimens for future molecular correlative studies.

X. To validate MAOA assessment in circulating tumor cells. XI. To assess correlation with tissue expression of MAOA. XII. To measure hypoxia-inducible factor (HIF)-1alpha expression and other potential biomarkers in circulating tumor cells as a potential measure of MAO activity.

TERTIARY OUTCOMES:

I. To measure expression of lysine-specific histone demethylase 1 (LSD1) in CRPC tumors that are progressing on docetaxel and correlate with the endpoints described in the primary objective and secondary objectives I, II, III, and V.

II. To conduct gene expression studies in CRPC tumors that are progressing on docetaxel and correlate them with and correlate with the endpoints described in the primary objective and secondary objectives I, II, III and V.

OUTLINE: This is a dose-escalation study of phenelzine sulfate.

Patients receive phenelzine sulfate orally (PO) once daily (QD) on days -7 to -4, and then twice daily (BID) on days -3 to 21. Patients receive docetaxel intravenously (IV) over 60 minutes on day 1. Treatment repeats every 21 days for at least 12 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of adenocarcinoma of the prostate
* Radiographic evidence of regional or distant metastases with suspected tumor in an area that is safe to biopsy
* Willingness to undergo tumor biopsy
* Evidence of CRPC indicated by history of progression despite standard hormonal therapy (by PSA and/or imaging studies)
* Planned or recent initiation of standard docetaxel therapy; patients may be enrolled after receiving standard docetaxel therapy as long as the patient has not demonstrated evidence of progression for more than 45 days before enrollment ("late enrollers")
* For patients who have been on anti-androgen therapy and had evidence of response to the addition of an anti-androgen (i.e., PSA reduction), patients must have discontinued anti-androgen therapy for at least six weeks (4 weeks for flutamide) without current evidence of an anti-androgen withdrawal response
* Serum testosterone levels < 50 ng/dL (unless surgically castrate); patients must continue androgen deprivation with an luteinizing hormone releasing hormone (LHRH) agonist if they have not undergone orchiectomy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Has recovered from all therapy-related toxicity to =< grade 2 (except alopecia, anemia and any signs or symptoms of androgen deprivation therapy)
* Absolute neutrophil count >= 1500/uL
* Platelets >= 100,000
* Creatinine =< 1.5 times upper limit of normal (ULN)
* Bilirubin =< 1.5 times ULN (if total bilirubin elevated, but direct is within normal limits [WNL], patient is eligible)
* Alanine aminotransferase (ALT) =< 2.5 times ULN
* PSA > 2 ng/mL (at the time of enrollment or prior to initiation of docetaxel)
* Life expectancy > 3 months
* Signed informed consent

Exclusion Criteria:

* Significant peripheral neuropathy defined as grade 2 or higher
* A second active malignancy except adequately treated non-melanoma skin cancer or other non-invasive or in situ neoplasm
* Significant active concurrent medical illness or infection precluding protocol treatment or survival
* Current uncontrolled hyperthyroidism
* Pheochromocytoma
* Carcinoid Syndrome
* Known or suspected brain metastases
* Treatment with radiotherapy within the past 4 weeks or radiopharmaceutical therapy (strontium, samarium) within the past 8 weeks
* Concurrent therapy with a Selective Serotonin Reuptake Inhibitor (SSRI), tricyclic antidepressant, or Monoamine Oxidase Inhibitor (MAOi); clinical judgment should be used in a decision to discontinue antidepressants; a minimum of a 1 week washout period is required for any tricyclic or related antidepressant, or any SSRI (2 weeks for paroxetine or sertraline, 5 weeks for fluoxetine); minimum 2 week washout for any MAOi
* Concurrent therapy with any excluded medications that cannot be safely discontinued prior to initiation of combination therapy; discontinuation prior to enrollment is not required, but discontinuation prior to combination therapy must be possible
* Caution should be exercised in patients who are regularly taking narcotic analgesics, particularly higher doses; the doses of narcotic analgesics may need to be reduced, patients may need to be monitored closely for drug interactions, and the risks and benefits of participation in the study should be considered; clinical judgment should be exercised to manage this potential drug interaction

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-07-12; Primary Completion 2016-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Beer, Principal Investigator — OHSU Knight Cancer Institute
Locations (3):
- United States (3):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Phenelzine and Docetaxel: Patients receive phenelzine sulfate orally (PO) once daily (QD) on days -7 to -4, and then twice daily (BID) on days -3 to 21. Patients receive docetaxel intravenously (IV) over 60 minutes on day 1. Treatment repeats every 21 days for at least 12 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Combination Phenelzine and Docetaxel
Started | 11
Completed | 6
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: 11 subjects received combination therapy
Groups:
- Combination Phenelzine and Docetaxel: Patients receive phenelzine sulfate PO QD on days -7 to -4, and then BID on days -3 to 21. Patients receive docetaxel IV over 60 minutes on day 1. Treatment repeats every 21 days for at least 12 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Combination Phenelzine and Docetaxel
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 68 [60 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Experience a PSA (Prostate-Specific Antigen) Decline of at Least 30%
Description: PSA response: A ≥ 30% reduction from baseline within 12 weeks of initiation of therapy (confirmed on a second measurement at least 3 weeks later).
Time Frame: Within 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Phenelzine and Docetaxel
Number analyzed (Participants) | 11
Participants | 2

2. Secondary Outcome: Duration of Progression Free Survival After Initiation of Combination Phenelzine and Docetaxel Therapy
Description: Progression free survival is calculated as the time from Day 1 of Combination therapy to first evidence of progression (by PSA, Measureable Disease, or Clinical Progression). For subjects who did not meet progression criteria, date of new therapy or date of death was used. Outcome is reported as mean.
Time Frame: Up to 6 years
Population: 1 subject withdrew from the study before the first evidence of progression and is not included in this progression free survival analysis.
Measure: Mean (Full Range); unit: days
Arm/Group | Combination Phenelzine and Docetaxel
Number analyzed (Participants) | 10
days | 77.9 [57 to 99]

3. Secondary Outcome: Frequency of MAOA (Monoamine Oxidase A) Overexpression in CRPC (Castration-Resistant Prostate Cancer) Tumors That Are Progressing on Docetaxel
Description: Reported as Number of participants with MAOA expression greater than 5%.
Time Frame: Baseline
Population: Subjects who had evaluable samples collected immediately prior to initiation of Combination Therapy. 3 subjects did not have evaluable samples and were not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Phenelzine and Docetaxel
Number analyzed (Participants) | 8
Participants | 8

4. Secondary Outcome: HIF-1alpha Expression in CTC (Circulating Tumor Cells) as a Potential Measure of MAO Activity
Time Frame: Up to 6 years
Population: Of eleven subjects, CTC samples were collected from only 3. No testing was conducted on these 3 samples.
Arm/Group | Combination Phenelzine and Docetaxel
Number analyzed (Participants) | 0

5. Secondary Outcome: MAOA Expression in CTC (Circulating Tumor Cells) and Comparison to Biopsy MAOA Expression
Description: A Pearson's correlation will be used to correlate tumor biopsy MAOA expression and circulating tumor cells MAOA expression.
Time Frame: Up to 6 years
Population: Of eleven subjects, CTC samples were collected from only 3. No testing was conducted on these 3 samples.
Arm/Group | Combination Phenelzine and Docetaxel
Number analyzed (Participants) | 0

6. Secondary Outcome: Maximum Change in PSA
Description: Measured from Day 1 of Combination therapy to PSA at 12 Weeks on therapy (or earlier if subject not on therapy for 12 weeks).
Time Frame: 12 weeks (or earlier in patients who discontinued early)
Population: 1 subject withdrew from the study before reaching 12 weeks and is not included in this progression free survival analysis.
Measure: Median (Full Range); unit: percentage of PSA change
Arm/Group | Combination Phenelzine and Docetaxel
Number analyzed (Participants) | 10
percentage of PSA change | 14.24 [-46.56 to 69.94]

7. Secondary Outcome: Response Rate in Measurable Disease by RECIST (Response Evaluation Criteria In Solid Tumors) Criteria
Description: Response in measurable disease is defined as a 30% decrease in the sum of diameters of target lesions (as described by RECIST 1.1).
Time Frame: Up to 6 years
Population: 3 subjects were excluded from this response rate calculation as they did not have additional scans beyond baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Phenelzine and Docetaxel
Number analyzed (Participants) | 8
Participants | 0

8. Secondary Outcome: Time to Death From All Causes
Description: Time to death is calculated from Day 1 of Combination therapy to death from any cause.
Time Frame: Up to 6 years
Measure: Median (Full Range); unit: days
Arm/Group | Combination Phenelzine and Docetaxel
Number analyzed (Participants) | 11
days | 191.0 [99 to 621]

9. Secondary Outcome: Toxicity of the Regimen
Description: Number of participants who experienced an Adverse Event. Detail of Adverse Events is reported in the Adverse Event Section
Time Frame: Up to 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Phenelzine and Docetaxel
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from start of Combination Therapy (phenelzine and docetaxel) until off study for progression, adverse event, or other reason.
Description: Serious Adverse Events are considered Serious only if they are both unexpected and related to study. Hospitalizations that are expected for these study agents or the study population are not considered Serious Adverse Events.
  Only Adverse Events that are considered possibly or definitely related to the study are reported.
Arm/Group | Combination Phenelzine and Docetaxel
All-Cause Mortality (participants affected / at risk) | 11/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Phenelzine and Docetaxel (N=11)
Sudden Death (General disorders) | 1 (11)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Phenelzine and Docetaxel (N=11)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
visual disturbance (Eye disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Edema (bilateral extremity) (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Thrush, oral (Infections and infestations) | 1 (1)
Weight gain (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain, back (Musculoskeletal and connective tissue disorders) | 1 (1)
Cyst, neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Concentration Impairment (Nervous system disorders) | 1 (1)
Sedation (Nervous system disorders) | 1 (1)
Pre-syncope (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Memory Loss (Nervous system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (torso) (Skin and subcutaneous tissue disorders) | 1 (1)
Nail Changes (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Hypertention (Vascular disorders) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed; overall morbidity of patient population prohibited long term treatment or follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes